CLINICAL TRIAL: NCT06930027
Title: Normobaric Hypoxia as a Strength Training Intensity Amplifier in Ice Hockey Players: Effects on Anaerobic Performance and Muscle Contraction Properties
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02/2024
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: High-intensity Strenght Training in Normoxia (H-N); Low-intensity Strenght Training in Normoxia (L-N); High-intensity Strenght Training in Normobaric Hypoxia (H-H); Low-intensity Strenght Training in Normobaric Hypoxia (L-H)
Keywords: resistance training; anaerobic performance; lactate clearance; muscle contractility; ice hockey; detraining prevention; injury rehabilitation
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High-intensity strength training under normoxic conditions (H-N) (Active Comparator): Participants performed supervised leg press resistance training twice weekly under normal oxygen conditions (normoxia, ~20.9% FiO₂). Each session consisted of four sets of 10 repetitions at 70-80% of their individual one-repetition maximum (1RM), progressively increasing from 70% (weeks 1-3) to 80% (weeks 4-6).
  Interventions: Other: Resistance Training (High-Intensity); Other: Normoxia
- Low-intensity strength training in normoxia (Active Comparator): Participants performed resistance training in normal oxygen conditions, using lower mechanical loads (20-30% 1RM) following a structured repetition scheme of 30/15/15/15 repetitions per session. Training intensity was progressively increased from 20% (weeks 1-3) to 30% (weeks 4-6).
  Interventions: Other: Resistance Training (High-Intensity); Other: Normoxia
- High-intensity strength training in hypoxia (Experimental): Participants conducted resistance training in normobaric hypoxia (simulated altitude ~3500 m; ~13.5% FiO₂), performing 4 sets × 10 repetitions at 70-80% 1RM, progressively increasing load from 70% (weeks 1-3) to 80% (weeks 4-6).
  Interventions: Other: Resistance Training (High-Intensity); Other: Normobaric Hypoxia
- Low-intensity strength training in hypoxia (Experimental): Participants completed resistance training in normobaric hypoxia (simulated altitude ~3500 m; ~13.5% FiO₂), employing a repetition scheme of 30/15/15/15 per session at 20-30% 1RM, with intensity progression from 20% (weeks 1-3) to 30% (weeks 4-6).
  Interventions: Other: Resistance Training (Low-Intensity); Other: Normobaric Hypoxia

INTERVENTIONS:
Other: Resistance Training (High-Intensity) — Leg press exercise performed at 70-80% of 1RM, structured as 4 sets × 10 repetitions, with controlled tempo and standardized rest intervals (2 minutes).
  Arms: High-intensity strength training in hypoxia; High-intensity strength training under normoxic conditions (H-N); Low-intensity strength training in normoxia
Other: Resistance Training (Low-Intensity) — Leg press exercise performed at 20-30% of 1RM, structured as 4 sets (30/15/15/15 repetitions), with controlled tempo and shorter rest intervals (1 minute).
  Arms: Low-intensity strength training in hypoxia
Other: Normobaric Hypoxia — Environmental intervention simulating an altitude of approximately 3500 meters (~13.5% FiO₂) using a normobaric hypoxic chamber.
  Arms: High-intensity strength training in hypoxia; Low-intensity strength training in hypoxia
Other: Normoxia — Training under normal atmospheric oxygen conditions (~20.9% FiO₂).
  Arms: High-intensity strength training under normoxic conditions (H-N); Low-intensity strength training in normoxia

SUMMARY:
The goal of this research study is to investigate the effects of resistance training performed under normobaric hypoxia (simulated altitude conditions) on anaerobic performance, lactate clearance, and muscle contractility in elite ice hockey players. The main questions it aims to answer are:

Does resistance training under hypoxic conditions improve anaerobic peak power and mean power compared to training under normal oxygen conditions?

Does training under hypoxia affect lactate kinetics and buffering capacity differently than normoxic training?

Does hypoxic training enhance muscle contractility properties differently compared to normoxic training?

In practice: Can hypoxic training help injured athletes maintain performance levels while reducing overall physical stress and preventing detraining?

Researchers will compare four training approaches:

High-intensity training in normoxia (normal oxygen conditions)

Low-intensity training in normoxia

High-intensity training in hypoxia (simulated altitude of 3500 meters)

Low-intensity training in hypoxia

Participants will:

Perform resistance training sessions using a leg press twice a week for 6 weeks, with progressively increased intensity.

Complete anaerobic performance tests (Wingate tests for both lower and upper limbs) before and after the training intervention.

Undergo tensiomyographic assessments to evaluate muscle contractility.

Provide capillary blood samples at 0, 4, and 8 minutes post-exercise to assess lactate clearance and metabolic recovery.

DETAILED DESCRIPTION:
Study Overview This study will investigate the physiological adaptations elicited by a structured resistance training program conducted under normobaric hypoxic conditions (simulated altitude of approximately 3500 meters) in comparison to normoxic training in elite ice hockey athletes. Specifically, the research will evaluate whether resistance training under hypoxic conditions can enhance anaerobic power output, accelerate lactate clearance kinetics, and positively influence muscle contractile properties. Furthermore, the study will examine the potential for hypoxic conditions to maintain or increase physiological training intensity while utilizing reduced mechanical loads, potentially lowering cumulative musculoskeletal stress. Additionally, the effectiveness of hypoxic training as a rehabilitation tool for injured athletes will be explored, assessing its capacity to preserve performance levels, facilitate recovery, and mitigate rapid detraining during periods of reduced training intensity.

Methods Participants Forty highly trained male ice hockey players will be recruited and randomly assigned to one of four experimental groups, with ten athletes per group (n = 10). All participants will provide written informed consent following a detailed explanation of the potential risks, benefits, and procedural requirements of the study. Inclusion criteria will stipulate that athletes have engaged in elite-level ice hockey training for at least three years and have no significant injury history within the preceding three months. Throughout the intervention period, participants will be instructed to maintain their habitual training routines, dietary practices, and recovery strategies to minimize potential confounding influences.

Study Design This investigation will be designed as a randomized controlled trial to compare the physiological effects of resistance training performed under normobaric hypoxia (simulated altitude equivalent to 3500 meters) versus normoxic conditions. Participants will be randomly allocated into one of four distinct intervention groups: (1) high-intensity training under normoxia (H-N), (2) low-intensity training under normoxia (L-N), (3) high-intensity training under hypoxia (H-H), and (4) low-intensity training under hypoxia (L-H). The training intervention will last six weeks, with each participant completing two supervised training sessions per week (totaling twelve sessions). Training adherence, technique consistency, and participant safety will be strictly monitored by experienced investigators throughout the study.

All training sessions will involve a standardized leg press exercise performed on identical equipment (a 45-degree plate-loaded leg press machine). Training loads, intensities, and repetition schemes will differ systematically based on group allocation. Athletes assigned to high-intensity training groups (H-N and H-H) will perform four sets of ten repetitions per session at 70-80% of their predetermined one-repetition maximum (1RM). Training load progression will be implemented systematically, beginning at 70% of 1RM during weeks 1-3 and increasing to 80% of 1RM during weeks 4-6. In contrast, athletes in low-intensity groups (L-N and L-H) will perform four sets per session using a repetition scheme of 30 repetitions in the first set, followed by three sets of 15 repetitions each (30/15/15/15), with loading progressing from 20% of 1RM in weeks 1-3 to 30% of 1RM in weeks 4-6.

All exercises will be executed with a controlled movement tempo (approximately two seconds for the eccentric phase and one second for the concentric phase). Rest periods will be standardized across groups: two minutes between sets for high-intensity groups and one minute between sets for low-intensity groups. Each session will begin with a standardized warm-up (five minutes of cycling at 100 W and one warm-up set at approximately 50% of the prescribed load) and conclude with a standardized cooldown (five minutes of cycling at 50 W). Load adjustments will be conducted weekly based on continuous monitoring to maintain the intended training intensity and progression.

Leg Press Protocol All resistance training sessions will be conducted using a standardized 45-degree plate-loaded leg press machine (Hammer Strength Linear Leg Press, Life Fitness, USA). Participants will execute the leg press exercise under strict supervision to ensure consistent technique, proper movement execution, and safety throughout the intervention.

Prior to initiating the training program, participants will complete a standardized one-repetition maximum (1RM) test on the leg press. This test will follow a structured incremental loading protocol with standardized rest intervals (3-5 minutes between attempts) and an adequate warm-up to ensure accurate baseline load determination.

Training sessions will be structured according to group allocation:

High-Intensity Training Groups (H-N and H-H):

In weeks 1-3, participants will perform four sets of ten repetitions at 70% of their individual 1RM. The load will be systematically increased to 80% of 1RM during weeks 4-6 while maintaining the same repetition scheme. Exercises will be executed with a controlled movement tempo (approximately two seconds for the eccentric phase and one second for the concentric phase), and rest intervals between sets will be standardized at two minutes.

Low-Intensity Training Groups (L-N and L-H):

In weeks 1-3, participants will complete four sets using a repetition scheme of 30 repetitions in the first set, followed by three sets of 15 repetitions each (30/15/15/15) at an intensity corresponding to 20% of their individual 1RM. The training load will be progressively increased to 30% of 1RM in weeks 4-6, using the same repetition scheme. Exercises will be conducted with the same controlled tempo (approximately two seconds for the eccentric phase and one second for the concentric phase) and standardized rest intervals of one minute between sets.

Each training session will begin with a standardized warm-up consisting of five minutes of cycling at 100 W, followed by one preparatory set on the leg press performed at approximately 50% of the planned training load. Sessions will conclude with a five-minute cooldown consisting of cycling at a low intensity (50 W). Training loads will be reviewed and adjusted weekly based on participant performance to ensure precise progression and maintenance of target intensities. Throughout each session, participants will receive continuous feedback regarding proper form, optimal range of motion (approximately 90° knee flexion at the deepest point), controlled breathing patterns, and consistent execution tempo.

Testing and Outcome Measures

Pre- and post-intervention assessments will be performed within one week before the commencement and one week after the completion of the six-week intervention period. The primary outcome measures will be as follows:

Anaerobic Performance:

Anaerobic power will be evaluated using Wingate Anaerobic Tests performed on a mechanically braked cycle ergometer (Monark 894E, Sweden). Participants will conduct two 30-second maximal effort tests for the lower limbs (separated by 20 minutes of passive recovery) to ensure reliability. An additional Wingate test for the upper limbs will be administered as an internal control measure. Both peak power (W) and mean power output (W) will be recorded and analyzed.

Lactate Kinetics and Buffering Capacity:

Lactate clearance will be assessed via capillary blood samples collected at baseline (immediately post-exercise, 0 minutes) and subsequently at 4 and 8 minutes post-exercise. Lactate concentrations (mmol·L-¹) will be analyzed using a validated portable lactate analyzer (Lactate Scout 4, EKF Diagnostics, Germany).

Muscle Contractility Assessment:

Muscle contractile properties will be assessed using tensiomyography (TMG) on two selected muscles: the vastus lateralis (the targeted muscle group involved in training) and the triceps brachii (an untrained control muscle). TMG measurements will include contraction time (Tc, ms) and maximal radial displacement (Dm, mm), which will provide insights into neuromuscular adaptations, muscle responsiveness, and contractile efficiency resulting from the intervention.

Statistical Analysis A priori sample size calculation will be conducted to ensure sufficient statistical power (β = 0.80) for detecting meaningful differences between groups. The analysis will indicate that a minimum of 10 participants per group (total N = 40) is required.

All statistical analyses will be performed using STATISTICA (TIBCO Software, USA) and GraphPad Prism version 10 (GraphPad Software, USA). Before inferential testing, data distributions will be evaluated for normality using the Shapiro-Wilk test, and variance homogeneity will be assessed with Levene's test. Descriptive statistics will be presented as means, standard deviations (SD), and 95% confidence intervals (CI).

A mixed-design split-plot ANOVA (2 × 4) will be employed to examine the main effects of Time (pre-intervention vs. post-intervention, within-subject factor), Group (H-N, L-N, H-H, L-H, between-subject factor), and the Time × Group interaction. The primary analytical focus will be on the interaction to determine if physiological adaptations in anaerobic performance, lactate clearance kinetics, and muscle contractile properties differ among the four training conditions.

Post-hoc analyses, using pairwise comparisons with Bonferroni adjustments, will be performed only in cases of significant interaction or main effects to pinpoint specific group differences. Descriptive statistics (means, standard deviations, and 95% confidence intervals) will be provided for clarity.

Effect sizes will be calculated as partial eta squared (η²) and interpreted according to Cohen's guidelines (small = 0.01-0.059, moderate = 0.06-0.137, large > 0.137). Outlier detection will be conducted systematically using box plots and Cook's distance to assess data quality and influential observations, with individual cases carefully evaluated and addressed if necessary.

Data normality and variance homogeneity assumptions will be verified using Shapiro-Wilk and Levene's tests, respectively. If these assumptions are violated, appropriate adjustments (such as Greenhouse-Geisser corrections) or non-parametric alternatives (e.g., Wilcoxon signed-rank or Friedman tests) will be applied. Additionally, regression analyses will be conducted to explore potential predictive relationships between physiological adaptations (lactate clearance and muscle contractile properties) and improvements in anaerobic performance measures.

Statistical significance will be interpreted as follows:

p < 0.05 will indicate moderate evidence against the null hypothesis, p < 0.01 will indicate strong evidence against the null hypothesis, p < 0.001 will represent very strong evidence against the null hypothesis. Outliers will be systematically identified using box plots and Cook's distance. Detected outliers will be individually reviewed to assess their impact and determine appropriate treatment (e.g., retention, exclusion, or sensitivity analysis).

Quality Assurance and Data Management Comprehensive Standard Operating Procedures (SOPs) will be developed and rigorously followed throughout the study. These SOPs will include explicit guidelines for participant recruitment procedures, informed consent acquisition, standardized data collection protocols, resistance training methodologies, lactate sampling techniques, tensiomyographic assessments, data entry and database management, adverse event identification and reporting, as well as measures to ensure data confidentiality and security.

Systematic data validation processes will be implemented regularly, assessing the completeness, accuracy, and internal consistency of recorded data. Automated range checks and logical consistency analyses will be embedded within the data management system, allowing for the immediate identification and correction of potential inconsistencies, inaccuracies, or protocol deviations.

Periodic source data verification audits will be conducted to ensure data accuracy and reliability. These audits will involve systematic cross-checking between electronic registry data and original source documents, including laboratory reports, electronic and paper-based case report forms, and raw physiological measurement outputs. This practice will ensure the fidelity and integrity of the recorded data.

A detailed data dictionary will be established, clearly defining all study variables. This dictionary will include descriptions of data coding schemes for categorical variables and physiological parameters, measurement units, calibration procedures of instruments, and reference physiological ranges applicable to each measurement. It will serve as a standardized reference tool to enhance data consistency and interpretability.

Missing data will be managed following predefined guidelines described explicitly in the study's statistical analysis plan. Strategies will include the exclusion of datasets with substantial missing data (i.e., more than 20% missing points per individual dataset) or the application of appropriate multiple-imputation techniques, depending on the nature and extent of the missing data. Sensitivity analyses will also be conducted to assess the robustness of study findings in response to different missing data treatments.

Finally, regular internal audits and continuous monitoring will be performed by the research team to verify adherence to the study protocols, data collection accuracy, participant compliance, and overall data integrity. Any identified deviations or irregularities will trigger immediate corrective actions, as detailed explicitly in the study's SOPs, thereby ensuring high-quality data collection and the validity and reliability of study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male professional-level ice hockey athletes (Napród Janów HC).
* Age range: 18-30 years.
* Minimum of 3 years of consistent professional level ice hockey training experience.
* No history of significant injury or illness within the previous 3 months.
* Able and willing to comply with all study procedures, including adherence to --scheduled training sessions and assessments.
* Provision of written informed consent to participate.

Exclusion Criteria:

* Current or recent (within past 3 months) musculoskeletal injuries or conditions that would limit participation in resistance training.
* Presence of cardiovascular, metabolic, respiratory, or neuromuscular disorders that may pose risk or interfere with performance assessment or training.
* Current participation in another structured hypoxic training protocol or simultaneous research intervention.
* History of altitude-related illness or known adverse reactions to hypoxic exposure.
* Use of any medications or supplements known to significantly influence muscular performance or recovery within four weeks prior to study initiation.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is restricted to participants who are biologically male and self-identify as male
Enrollment: 40 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Anaerobic Performance (2x Wingate Test) | Baseline (pre-intervention) and 6 weeks (immediately post-intervention)
  Change in anaerobic performance will be assessed using peak power (W) and mean power output (W), determined through the Wingate Anaerobic Test performed on a cycle ergometer. Lower-limb anaerobic performance will be evaluated by two consecutive Wingate tests, separated by a 20-minute rest period, to ensure reliability. An additional Wingate test for the upper limbs serves as an internal control.
Lactate Clearance Kinetics | Baseline (pre-intervention) and 6 weeks (post-intervention)
  Capillary blood lactate concentrations will be assessed at baseline (0 min immediately post-exercise), and at 4 and 8 minutes post-exercise, to evaluate lactate production and clearance kinetics following maximal anaerobic efforts.
Muscle Contractility (Tensiomyography) | Time Frame: Baseline (pre-intervention) and 6 weeks (post-intervention)
  Muscle contractile properties (contraction time-Tc, and maximal radial displacement-Dm) will be assessed via tensiomyography (TMG) on the vastus lateralis muscle (trained muscle group) and triceps brachii (untrained control muscle), to evaluate neuromuscular adaptations following the intervention.

SECONDARY OUTCOMES:
Maximal Strength (1-Repetition Maximum, 1RM) | Baseline (pre-intervention) and 6 weeks (immediately post-intervention)
  Maximal lower limb strength will be assessed by determining participants' one-repetition maximum (1RM) on the leg press exercise. The test will be performed following standardized incremental loading protocols, including appropriate rest intervals and warm-up procedures. Changes in maximal strength will indicate muscular adaptation resulting from the training interventions.

OTHER OUTCOMES:
Perceived Effort and Fatigue (Rating of Perceived Exertion - RPE) | Recorded twice weekly, during all training sessions over the 6-week intervention (weeks 1-6).
  Participants' subjective perception of effort and fatigue will be monitored using a validated Rating of Perceived Exertion (RPE) scale (, Borg CR-10). RPE will be recorded immediately following each set during training sessions to quantify subjective training intensity and track fatigue progression across the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Jerzy Kukuczka Academy of Physical Education in Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Data collected during this study will be available upon reasonable request. Individual participant data sharing will be considered on a case-by-case basis, subject to ethical approval, participant consent, and data protection regulations. Data requests must clearly outline the purpose, intended analyses, and measures taken to ensure confidentiality and data security.